CLINICAL TRIAL: NCT00315302
Title: A Randomized Trial Comparing Atropine to Atropine Plus a Plano Lens for the Sound Eye As Prescribed Treatments for Amblyopia in Children 3 to <7 Years Old
Brief Title: Trial Comparing Atropine to Atropine Plus a Plano Lens for the Sound Eye for Amblyopia in Children 3 to <7 Years Old
Acronym: ATS8
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Ray Kraker, Director, PEDIG Coordinating Center, Jaeb Center for Health Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEI-115; 2U10EY011751 (NIH)
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Amblyopia
Keywords: Amblyopia; Atropine; Plano lens
MeSH Terms: conditions — Amblyopia | interventions — Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atropine (Active Comparator): Atropine 1% once each weekend day in the sound eye
  Interventions: Drug: Atropine
- Atropine plus plano (Active Comparator): Atropine 1% once each weekend day in the sound eye plus a plano lens for the sound eye
  Interventions: Drug: Atropine; Device: Plano Lens

INTERVENTIONS:
Drug: Atropine — Atropine 1% once each weekend day
Device: Plano Lens — Plano lens for the sound eye
  Arms: Atropine plus plano

SUMMARY:
The purpose of the study is:

* To compare the effectiveness and safety of weekend atropine augmented with a plano lens for the sound eye versus weekend atropine alone for moderate amblyopia (20/40 to 20/100) in children 3 to less than 7 years old.
* To provide data on the response of severe amblyopia (20/125 to 20/400) to atropine treatment with and without a plano lens.

DETAILED DESCRIPTION:
Atropine is an effective treatment of moderate amblyopia. Reduction of the plus sphere for the sound eye is an accepted method of enhancing and possibly accelerating the treatment effect. Demonstrating additional value of the plano lens in terms of speed of improvement will shorten the treatment period, possibly improving child and parental compliance, leading to improved overall outcomes for patients with amblyopia. If the plano lens leads to greater improvement, then there will be less permanent visual impairment in patients with a history of amblyopia. It also is important to determine if the use of a plano lens in conjunction with atropine has a deleterious effect on the sound eye, and if yes, how often this occurs.

Little is known about the pharmacologic treatment of severe amblyopia. This study will provide important prospectively determined outcome data at little additional expense.

In a study conducted by the Pediatric Eye Disease Investigator Group, A Randomized Trial Comparing Daily Atropine Versus Weekend Atropine for Moderate Amblyopia, the use of weekend atropine for moderate amblyopia was as effective as daily treatment. Intermittent atropine use (such as using it only on the weekends) has the theoretical potential benefit of the sound eye having some time each week during which cycloplegia is only partial. It is possible that allowing some loss of the cycloplegic effect over the course of each week may be safer for the sound eye.

The study has been designed as a simple trial that, other than the type of amblyopia therapy being determined through the randomization process, approximates standard clinical practice. The two treatment regimes for the 18 week primary treatment period are: 1) Atropine 1% once each weekend day in the sound eye and 2) Atropine 1% once each weekend day in the sound eye plus a plano lens for the sound eye.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 3 to less than 7 years old with amblyopia associated with strabismus, anisometropia, or both.
* Visual acuity in the amblyopic eye must be between 20/40 and 20/400 inclusive, visual acuity in the sound eye 20/40 or better and inter-eye acuity difference > 3 logMAR lines.
* Spectacles, if needed, must be worn for at least 16 weeks or until visual acuity documented to be stable.

Exclusion Criteria:

* Atropine treatment within 6 months of enrollment and other amblyopia treatment of any type (other than normal spectacle lenses) used within one month of enrollment
* No myopia in amblyopic eye

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2005-02; Primary Completion 2007-10 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Weakley, M.D., Study Chair — University of Texas Southwestern Medical Center; Susan A. Cotter, O.D., Study Chair — Southern California College of Optometry at Marshall B. Ketchum University
Locations (2):
- United States (2):
  - Southern California College of Optometry, Fullerton, California
  - UT Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Result] Pediatric Eye Disease Investigator Group. Pharmacological plus optical penalization treatment for amblyopia: results of a randomized trial. Arch Ophthalmol. 2009 Jan;127(1):22-30. doi: 10.1001/archophthalmol.2008.520. PMID 19139333
- [Result] Repka MX, Kraker RT, Beck RW, Birch E, Cotter SA, Holmes JM, Hertle RW, Hoover DL, Klimek DL, Marsh-Tootle W, Scheiman MM, Suh DW, Weakley DR; Pediatric Eye Disease Investigator Group. Treatment of severe amblyopia with weekend atropine: results from 2 randomized clinical trials. J AAPOS. 2009 Jun;13(3):258-63. doi: 10.1016/j.jaapos.2009.03.002. PMID 19541265
- [Derived] Wallace DK, Lazar EL, Melia M, Birch EE, Holmes JM, Hopkins KB, Kraker RT, Kulp MT, Pang Y, Repka MX, Tamkins SM, Weise KK; Pediatric Eye Disease Investigator Group. Stereoacuity in children with anisometropic amblyopia. J AAPOS. 2011 Oct;15(5):455-61. doi: 10.1016/j.jaapos.2011.06.007. PMID 22108357
- [Derived] Repka M, Simons K, Kraker R; Pediatric Eye Disease Investigator Group. Laterality of amblyopia. Am J Ophthalmol. 2010 Aug;150(2):270-4. doi: 10.1016/j.ajo.2010.01.040. Epub 2010 May 8. PMID 20451898

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between Feb 2005 and May 2007, 240 subjects were randomized at 30 sites (180 with moderate amblyopia 20/40 to 20/100 in a primary cohort, and an additional 60 with severe amblyopia 20/125 to 20/400 that were followed as a secondary cohort).
Pre-assignment Details: Subjects must have had stable visual acuity in glasses (if applicable) before enrollment and randomization.
Groups:
- Atropine-Moderate Amblyopia: Atropine 1% once each weekend day in the sound eye among patients with moderate amblyopia (20/40 to 20/100)
- Atropine Plus Plano-Moderate Amblyopia: Atropine 1% once each weekend day in the sound eye plus a plano lens for the sound eye among patients with moderate amblyopia (20/40 to 20/100)
- Atropine-Severe Amblyopia: Atropine 1% once each weekend day in the sound eye among patients with severe (20/125 to 20/400)
- Atropine Plus Plano-Severe Amblyopia: Atropine 1% once each weekend day in the sound eye plus a plano lens for the sound eye among patients with severe amblyopia (20/125 to 20/400)
Period: Overall Study
Arm/Group | Atropine-Moderate Amblyopia | Atropine Plus Plano-Moderate Amblyopia | Atropine-Severe Amblyopia | Atropine Plus Plano-Severe Amblyopia
Started | 90 | 90 | 26 | 34
5 Week Visit | 85 | 86 | 26 | 30
10 Week Visit | 86 (Can be higher as includes subjects who may have missed the 5 week visit) | 85 | 24 | 29
18 Week Primary Outcome Visit | 84 | 88 (Can be higher as includes subjects who may have missed the 10 week or other visit) | 24 | 31 (Can be higher as includes subjects who may have missed the 10 week or other visit)
Partial Responder Phase (Post 18 Weeks) | 16 (Those who improved in the amblyopic eye at 18wk outcome continued on treatment w/ visits every 8wks.) | 13 (Those who improved in the amblyopic eye at 18wk outcome continued on treatment w/ visits every 8wks.) | 9 (Those who improved in the amblyopic eye at 18wk outcome continued on treatment w/ visits every 8wks.) | 11 (Those who improved in the amblyopic eye at 18wk outcome continued on treatment w/ visits every 8wks.)
Completed | 84 (Completed defined as completing 18 week primary outcome exam) | 88 (Completed defined as completing 18 week primary outcome exam) | 24 (Completed defined as completing 18 week primary outcome exam) | 31 (Completed defined as completing 18 week primary outcome exam)
Not Completed | 6 | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atropine-Moderate Amblyopia | Atropine Plus Plano-Moderate Amblyopia | Atropine-Severe Amblyopia | Atropine Plus Plano-Severe Amblyopia | Total
Number analyzed (Participants) | 90 | 90 | 26 | 34 | 240
Age, Categorical [Count of Participants; unit: Participants] — Age at enrollment
  Participants
    <=18 years | 90 | 90 | 26 | 34 | 240
    Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
    >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at enrollment
  years | 5.2 (1.1) | 5.1 (1.0) | 4.5 (0.9) | 4.4 (1.0) | 5.0 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 47 | 8 | 16 | 118
  Male | 43 | 43 | 18 | 18 | 122
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 75 | 70 | 23 | 28 | 196
  African-American | 1 | 4 | 1 | 3 | 9
  Hispanic or Latino | 12 | 14 | 2 | 3 | 31
  Asian | 1 | 2 | 0 | 0 | 3
  Unknown / Not reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 89 | 90 | 26 | 34 | 239
  Canada | 1 | 0 | 0 | 0 | 1
Cause of Amblyopia [Number; unit: participants]
  Strabismus | 38 | 37 | 10 | 11 | 96
  Anisometropia | 32 | 30 | 5 | 8 | 75
  Strabismus and anisometropia | 20 | 23 | 11 | 15 | 69
Distance Visual Acuity in Amblyopic Eye [Number; unit: participants] — Visual acuity is measured in each eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol at 18 weeks resulting in a Snellen acuity score that can range from 20/16 to 20/800. This visual acuity score is converted to logMAR (log of min angle of resolution) for statistical analysis.
  20/16=-0.1 logMAR; best 20/20=0.0 logMAR; 20/25=0.1; 20/32=0.2; 20/40=0.3; 20/50=0.4; 20/63=0.5; 20/80=0.6; 20/100=0.7; 20/125=0.8; 20/160=0.9; 20/200=1.0; 20/250=1.1; 20/320=1.2; 20/400=1.3; 20/500=1.4; 20/640=1.5; 20/800=1.6; worst
  participants
    20/400 (worse) | 0 | 0 | 0 | 8 | 8
    20/320 | 0 | 0 | 8 | 2 | 10
    20/250 | 0 | 0 | 1 | 3 | 4
    20/200 | 0 | 0 | 5 | 5 | 10
    20/160 | 0 | 0 | 5 | 5 | 10
    20/125 | 0 | 0 | 7 | 11 | 18
    20/100 | 7 | 15 | 0 | 0 | 22
    20/80 | 14 | 15 | 0 | 0 | 29
    20/63 | 29 | 28 | 0 | 0 | 57
    20/50 | 24 | 17 | 0 | 0 | 41
    20/40 (better) | 16 | 15 | 0 | 0 | 31
Distance Visual Acuity in Sound Eye [Number; unit: participants] — Visual acuity is measured in each eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol at 18 weeks resulting in a Snellen acuity score that can range from 20/16 to 20/800. This visual acuity score is converted to logMAR (log of min angle of resolution) for statistical analysis.
  20/16=-0.1 logMAR; best 20/20=0.0 logMAR; 20/25=0.1; 20/32=0.2; 20/40=0.3; 20/50=0.4; 20/63=0.5; 20/80=0.6; 20/100=0.7; 20/125=0.8; 20/160=0.9; 20/200=1.0; 20/250=1.1; 20/320=1.2; 20/400=1.3; 20/500=1.4; 20/640=1.5; 20/800=1.6; worst
  participants
    20/40 (worse) | 3 | 3 | 4 | 7 | 17
    20/32 | 18 | 18 | 11 | 12 | 59
    20/25 | 27 | 28 | 8 | 7 | 70
    20/20 | 31 | 33 | 3 | 8 | 75
    20/16 (better) | 11 | 8 | 0 | 0 | 19
Prior Treatment for Amblyopia at Enrollment [Number; unit: participants]
  None | 76 | 72 | 24 | 28 | 200
  Patching | 9 | 12 | 1 | 6 | 28
  Atropine | 1 | 2 | 0 | 0 | 3
  Patching and Atropine | 4 | 4 | 1 | 0 | 9
Refractive Error in Amblyopic Eye (spherical equivalent/diopters) [Number; unit: participants] — Measured in diopters (D) using cycloplegic refraction sphere, cylinder, and axis. Spherical equivalent is defined as the sphere plus 1/2 the cylinder.
  participants
    0 to < +1.00 D | 1 | 0 | 0 | 0 | 1
    +1.00 to < +2.00 D | 0 | 6 | 1 | 0 | 7
    +2.00 D to < +3.00 D | 8 | 6 | 3 | 0 | 17
    +3.00 D to < +4.00 D | 13 | 15 | 3 | 4 | 35
    >= +4.00 D | 68 | 63 | 19 | 30 | 180
Refractive Error in Sound Eye (spherical equivalent/diopters) [Number; unit: participants] — Measured in diopters (D) using cycloplegic refraction sphere, cylinder, and axis. Spherical equivalent is defined as the sphere plus 1/2 the cylinder.
  participants
    + 1.50 to < + 2.00 D | 17 | 23 | 6 | 6 | 52
    + 2.00 D to < + 3.00 D | 14 | 19 | 8 | 5 | 46
    +3.00 D to < + 4.00 D | 20 | 12 | 2 | 8 | 42
    >= + 4.00 D | 39 | 36 | 10 | 15 | 100
Distance Visual Acuity in Amblyopic Eye [Mean (Standard Deviation); unit: log of min angle of resolution (logMAR)] — Visual acuity is measured in each eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol at 18 weeks resulting in a Snellen acuity score that can range from 20/16 to 20/800. This visual acuity score is converted to logMAR (log of min angle of resolution) for statistical analysis.
  20/16=-0.1 logMAR; best 20/20=0.0 logMAR; 20/25=0.1; 20/32=0.2; 20/40=0.3; 20/50=0.4; 20/63=0.5; 20/80=0.6; 20/100=0.7; 20/125=0.8; 20/160=0.9; 20/200=1.0; 20/250=1.1; 20/320=1.2; 20/400=1.3; 20/500=1.4; 20/640=1.5; 20/800=1.6; worst
  log of min angle of resolution (logMAR) | 0.47 (0.12) | 0.50 (0.13) | 0.99 (0.16) | 1.01 (0.20) | 0.61 (0.27)
Distance Visual Acuity in Sound Eye [Mean (Standard Deviation); unit: log of min angle of resolution (logMAR)] — Visual acuity is measured in each eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol at 18 weeks resulting in a Snellen acuity score that can range from 20/16 to 20/800. This visual acuity score is converted to logMAR (log of min angle of resolution) for statistical analysis.
  20/16=-0.1 logMAR; best 20/20=0.0 logMAR; 20/25=0.1; 20/32=0.2; 20/40=0.3; 20/50=0.4; 20/63=0.5; 20/80=0.6; 20/100=0.7; 20/125=0.8; 20/160=0.9; 20/200=1.0; 20/250=1.1; 20/320=1.2; 20/400=1.3; 20/500=1.4; 20/640=1.5; 20/800=1.6; worst
  log of min angle of resolution (logMAR) | 0.07 (0.10) | 0.07 (0.10) | 0.16 (0.09) | 0.15 (0.11) | .09 (.11)
Intereye Acuity Difference [Mean (Standard Deviation); unit: logMAR lines] — Intereye difference defined as the difference between logMAR scores (amblyopic eye minus sound eye)
  logMAR lines | 4.0 (1.2) | 4.3 (1.3) | 8.3 (1.7) | 8.6 (2.2) | 5.2 (2.4)
Refractive Error in Amblyopic Eye (spherical equivalent/diopters) [Mean (Standard Deviation); unit: diopters] — Measured in diopters (D) using cycloplegic refraction sphere, cylinder, and axis. Spherical equivalent is defined as the sphere plus 1/2 the cylinder.
  diopters | 4.99 (1.66) | 4.94 (1.81) | 5.25 (2.09) | 5.36 (1.29) | 5.05 (1.72)
Refractive Error in Sound Eye (spherical equivalent/diopters) [Mean (Standard Deviation); unit: diopters] — Measured in diopters (D) using cycloplegic refraction sphere, cylinder, and axis. Spherical equivalent is defined as the sphere plus 1/2 the cylinder.
  diopters | 3.71 (1.71) | 3.54 (1.86) | 3.60 (2.18) | 3.71 (1.58) | 3.63 (1.79)

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity Mean Score in the Amblyopic Eye
Description: Visual acuity is measured in each eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol at 18 weeks resulting in an Snellen equivalent acuity score that can range from 20/16 to 20/800. This visual acuity score is converted to logMAR (log of min angle of resolution) for statistical analysis.
  20/16=-0.1 logMAR; best 20/20=0.0 logMAR; 20/25=0.1; 20/32=0.2; 20/40=0.3; 20/50=0.4; 20/63=0.5; 20/80=0.6; 20/100=0.7; 20/125=0.8; 20/160=0.9; 20/200=1.0; 20/250=1.1; 20/320=1.2; 20/400=1.3; 20/500=1.4; 20/640=1.5; 20/800=1.6; worst
Time Frame: 18 weeks
Population: Primary analysis includes only patients who completed the 18 week exam. No imputation was done if missed exam; analysis followed the intent to treat principle.
Measure: Mean (Standard Deviation); unit: logMAR units
Arm/Group | Atropine-Moderate Amblyopia | Atropine Plus Plano-Moderate Amblyopia | Atropine-Severe Amblyopia | Atropine Plus Plano-Severe Amblyopia
Number analyzed (Participants) | 84 | 88 | 24 | 31
logMAR units | 0.23 (0.16) | 0.22 (0.20) | 0.54 (0.26) | 0.50 (0.38)
Statistical Analysis 1: Comparison: Atropine-Moderate Amblyopia vs Atropine Plus Plano-Moderate Amblyopia; The primary analysis was a treatment group comparison of logMAR visual acuity scores in the amblyopic eye obtained 18 weeks after randomization, adjusted for baseline acuity scores in an analysis of covariance (ANCOVA) model. The primary analysis included only patients with visual acuity of 20/40 to 20/100; sample size was based upon a two-sided alpha of 0.05, with 90% power to detect a difference if the true difference in change from baseline between groups was 0.075 logMAR at 18 weeks; Test type: Superiority or Other; p = 0.21, ANCOVA; Mean Difference (Final Values) = 0.3, 95% CI [-0.2 to 0.8], Standard Deviation 0.24 — The difference was calculated as atropine plus plano group minus atropine group

2. Primary Outcome: Visual Acuity Distribution in the Amblyopic Eye
Description: Visual acuity is measured in each eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol at 18 weeks resulting in a Snellen acuity score that can range from 20/16 to 20/800. This visual acuity score is converted to logMAR (log of min angle of resolution) for statistical analysis.
  20/16=-0.1 logMAR; best 20/20=0.0 logMAR; 20/25=0.1; 20/32=0.2; 20/40=0.3; 20/50=0.4; 20/63=0.5; 20/80=0.6; 20/100=0.7; 20/125=0.8; 20/160=0.9; 20/200=1.0; 20/250=1.1; 20/320=1.2; 20/400=1.3; 20/500=1.4; 20/640=1.5; 20/800=1.6; worst
Time Frame: 18 weeks
Measure: Number; unit: Participants
Arm/Group | Atropine-Moderate Amblyopia | Atropine Plus Plano-Moderate Amblyopia | Atropine-Severe Amblyopia | Atropine Plus Plano-Severe Amblyopia
Number analyzed (Participants) | 84 | 88 | 24 | 31
Participants
  20/400 (worse) | 0 | 0 | 0 | 1
  20/320 | 0 | 0 | 0 | 1
  20/250 | 0 | 0 | 1 | 2
  20/200 | 0 | 0 | 0 | 0
  20/160 | 0 | 1 | 2 | 1
  20/125 | 0 | 1 | 4 | 4
  20/100 | 2 | 1 | 1 | 2
  20/80 | 2 | 4 | 1 | 2
  20/63 | 4 | 6 | 5 | 2
  20/50 | 6 | 7 | 5 | 4
  20/40 | 18 | 9 | 3 | 0
  20/32 | 28 | 24 | 1 | 8
  20/25 | 12 | 19 | 0 | 1
  20/20 | 11 | 12 | 1 | 1
  20/16 (better) | 1 | 4 | 0 | 2
Statistical Analysis 1: Comparison: Atropine-Moderate Amblyopia vs Atropine Plus Plano-Moderate Amblyopia; Null hypothesis: proportion 20/25 or better at 18wks in atropine group = proportion 20/25 or better at 18wks in atropine plus plano group Alternative hypothesis: proportion 20/25 or better at 18wks in atropine group NOT equal to proportion 20/25 or better at 18wks in atropine plus plano group; Test type: Superiority or Other; p = .03, Regression, Logistic; proportion 20/25 as a function of treatment group controlling for baseline acuity

3. Primary Outcome: Mean Change in Visual Acuity in the Amblyopic Eye
Description: Acuity is measured in each eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol at baseline and at 18wks resulting in a Snellen acuity score that can range from 20/16 to 20/800. The score is converted to logMAR (log of min angle of resolution) for statistical analysis, and a difference between the scores is calculated.
  A positive difference indicates acuity was better at 18wks than at baseline; a negative difference indicates acuity was worse at 18wks than at baseline.
Time Frame: baseline to 18 weeks
Measure: Mean (Standard Deviation); unit: logMAR units
Arm/Group | Atropine-Moderate Amblyopia | Atropine Plus Plano-Moderate Amblyopia | Atropine-Severe Amblyopia | Atropine Plus Plano-Severe Amblyopia
Number analyzed (Participants) | 84 | 88 | 24 | 31
logMAR units | 2.4 (1.4) | 2.8 (1.8) | 4.5 (3.1) | 5.1 (3.7)
Statistical Analysis 1: Comparison: Atropine-Severe Amblyopia; 95% confidence interval calculated within treatment group on the amount of change from baseline; Test type: Superiority or Other; Mean Difference (Final Values) = 4.5, 95% CI 2-sided [3.2 to 5.8], Standard Deviation 3.1
Statistical Analysis 2: Comparison: Atropine Plus Plano-Severe Amblyopia; 95% confidence interval calculated within treatment group on the amount of change from baseline; Test type: Superiority or Other; Mean Difference (Final Values) = 5.1, 95% CI 2-sided [3.7 to 6.4], Standard Deviation 3.7

4. Primary Outcome: Distribution of Change in Visual Acuity in the Amblyopic Eye
Description: as for outcome 3
Time Frame: baseline to 18 weeks
Measure: Number; unit: Participants
Arm/Group | Atropine-Moderate Amblyopia | Atropine Plus Plano-Moderate Amblyopia | Atropine-Severe Amblyopia | Atropine Plus Plano-Severe Amblyopia
Number analyzed (Participants) | 84 | 88 | 24 | 31
Participants
  -3 (worse) | 0 | 1 | 0 | 0
  -2 | 0 | 0 | 0 | 1
  -1 | 2 | 2 | 0 | 1
  0 | 4 | 5 | 2 | 2
  +1 | 18 | 11 | 2 | 3
  +2 | 18 | 19 | 3 | 1
  +3 | 22 | 18 | 3 | 2
  +4 | 17 | 18 | 4 | 3
  >= +5 (better) | 3 | 14 | 3 | 3
Statistical Analysis 1: Comparison: Atropine-Moderate Amblyopia vs Atropine Plus Plano-Moderate Amblyopia; Null hypothesis: proportion 3 or more lines better at 18wks in atropine group = proportion 3 or more lines better at 18wks in atropine plus plano group Alternative hypothesis: proportion 3 or more lines better at 18wks in atropine group NOT equal to proportion 3 or more lines better at 18wks in atropine plus plano group; Test type: Superiority or Other; p = 0.39, Regression, Logistic; proportion 20/25 as a function of treatment group controlling for baseline acuity

5. Secondary Outcome: Randot Preschool Stereoacuity at 18 Weeks- Participants With All Causes of Amblyopia
Description: The Randot Preschool Stereotest measures stereopsis from 800 to 40 seconds of arc on patients as young as 2 years of age. This Stereotest is designed as a matching game in which the patient matches pictures in a test booklet wearing special glasses. A subject can fail the pretest (not see any pictures) or can score >800 (the worst), 800, 400, 200, 100, 60, or 40 (the best) seconds of arc. If two shapes are identified correctly the patient progresses to the next lower stereoacuity level. A failed test occurs when the patient cannot identify any shapes.
Time Frame: 18 weeks
Population: Not reported among subjects with severe amblyopia
Measure: Number; unit: Participants
Arm/Group | Atropine-Moderate Amblyopia | Atropine Plus Plano-Moderate Amblyopia | Atropine-Severe Amblyopia | Atropine Plus Plano-Severe Amblyopia
Number analyzed (Participants) | 84 | 88 | 0 | 0
Participants
  Failed black & white shape identification pretest | 3 | 4 |  |
  >800 arcsec (worst) | 40 | 41 |  |
  800 arcsec | 7 | 10 |  |
  400 arcsec | 11 | 12 |  |
  200 arcsec | 10 | 6 |  |
  100 arcsec | 4 | 10 |  |
  60 arcsec | 5 | 1 |  |
  40 arcsec (best) | 2 | 1 |  |
  Not done | 2 | 3 |  |
Statistical Analysis 1: Comparison: Atropine-Moderate Amblyopia vs Atropine Plus Plano-Moderate Amblyopia; All patients without respect to cause of amblyopia; Test type: Superiority or Other; p = 0.39, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test to evaluate difference in change from baseline in stereoacuity by treatment group

6. Secondary Outcome: Randot Preschool Stereoacuity at 18 Weeks- Anisometropic Participants Only
Description: as for outcome 5
Time Frame: 18 weeks
Population: Not reported among subjects with severe amblyopia
Measure: Number; unit: Participants
Arm/Group | Atropine-Moderate Amblyopia | Atropine Plus Plano-Moderate Amblyopia | Atropine-Severe Amblyopia | Atropine Plus Plano-Severe Amblyopia
Number analyzed (Participants) | 29 | 30 | 0 | 0
Participants
  Failed black & white shape identification pretest | 0 | 0 |  |
  >800 arcsec (worst) | 7 | 9 |  |
  800 arcsec | 2 | 3 |  |
  400 arcsec | 5 | 6 |  |
  200 arcsec | 8 | 3 |  |
  100 arcsec | 3 | 6 |  |
  60 arcsec | 1 | 1 |  |
  40 arcsec (best) | 2 | 1 |  |
  Not done | 1 | 1 |  |
Statistical Analysis 1: Comparison: Atropine-Moderate Amblyopia vs Atropine Plus Plano-Moderate Amblyopia; Among anisometropic patients only; Test type: Superiority or Other; p = 0.90, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test to evaluate difference in change from baseline in stereoacuity by treatment group

7. Secondary Outcome: Mean Change in Visual Acuity in the Sound Eye
Description: as for outcome 3
Time Frame: baseline to 18 weeks
Measure: Mean (Standard Deviation); unit: logMAR units
Arm/Group | Atropine-Moderate Amblyopia | Atropine Plus Plano-Moderate Amblyopia | Atropine-Severe Amblyopia | Atropine Plus Plano-Severe Amblyopia
Number analyzed (Participants) | 84 | 88 | 24 | 31
logMAR units | 0.4 (0.9) | 0.0 (1.0) | 0.10 (0.12) | 0.15 (0.15)

8. Secondary Outcome: Distribution of Change in Visual Acuity in the Sound Eye
Description: as for outcome 3
Time Frame: baseline to 18 weeks
Measure: Number; unit: Participants
Arm/Group | Atropine-Moderate Amblyopia | Atropine Plus Plano-Moderate Amblyopia | Atropine-Severe Amblyopia | Atropine Plus Plano-Severe Amblyopia
Number analyzed (Participants) | 84 | 88 | 24 | 31
Participants
  -4 (worse) | 1 | 1 | 0 | 0
  -3 | 0 | 1 | 0 | 0
  -2 | 0 | 3 | 1 | 4
  -1 | 3 | 12 | 0 | 2
  0 | 49 | 50 | 11 | 13
  +1 | 24 | 17 | 9 | 12
  +2 | 6 | 4 | 3 | 0
  +3 (better) | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Atropine-Moderate Amblyopia vs Atropine Plus Plano-Moderate Amblyopia; Null hypothesis: proportion 1 or more lines worse and worse than 20/20 at 18wks same in both groups; Alternate: proportion 1 or more lines worse and worse than 20/20 at 18wks same in both groups; Test type: Superiority or Other; p = 0.003, Fisher Exact

9. Secondary Outcome: Visual Acuity Distribution in the Sound Eye
Description: Acuity is measured in each eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol at baseline and at 18 wks resulting in a Snellen acuity score that can range from 20/16 to 20/800. This acuity score is converted to logMAR (log of min angle of resolution) for statistical analysis.
  20/16=-0.1 logMAR; best 20/20=0.0 logMAR; 20/25=0.1; 20/32=0.2; 20/40=0.3; 20/50=0.4; 20/63=0.5; 20/80=0.6; 20/100=0.7; 20/125=0.8; 20/160=0.9; 20/200=1.0; 20/250=1.1; 20/320=1.2; 20/400=1.3; 20/500=1.4; 20/640=1.5; 20/800=1.6; worst
Time Frame: 18 weeks
Measure: Number; unit: Participants
Arm/Group | Atropine-Moderate Amblyopia | Atropine Plus Plano-Moderate Amblyopia | Atropine-Severe Amblyopia | Atropine Plus Plano-Severe Amblyopia
Number analyzed (Participants) | 84 | 88 | 24 | 31
Participants
  20/63 (worse) | 1 | 1 | 0 | 1
  20/50 | 0 | 3 | 1 | 3
  20/40 | 2 | 3 | 1 | 4
  20/32 | 10 | 16 | 6 | 7
  20/25 | 14 | 22 | 8 | 7
  20/20 | 36 | 28 | 6 | 7
  20/16 (better) | 21 | 15 | 2 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the 18wk outcome visit.
Arm/Group | Atropine-Moderate Amblyopia | Atropine Plus Plano-Moderate Amblyopia | Atropine-Severe Amblyopia | Atropine Plus Plano-Severe Amblyopia
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/90 | 0/26 | 0/34
Other Adverse Events (participants affected / at risk) | 8/90 | 1/90 | 1/26 | 5/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atropine-Moderate Amblyopia (N=90) | Atropine Plus Plano-Moderate Amblyopia (N=90) | Atropine-Severe Amblyopia (N=26) | Atropine Plus Plano-Severe Amblyopia (N=34)
Light sensitivity (Eye disorders) | 8 (8) | 1 (1) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No